CLINICAL TRIAL: NCT02832557
Title: Validation of a Salivary miRNA Diagnostic Test for Autism Spectrum Disorder
Brief Title: A Salivary miRNA Diagnostic Test for Autism
Status: Completed | Type: Observational
Sponsor: State University of New York - Upstate Medical University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Quadrant Biosciences Inc. (Industry); Milton S. Hershey Medical Center (Other); University of Missouri-Columbia (Other); Children's Hospital Medical Center, Cincinnati (Other); Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Frank A Middleton, Principal Investigator/Associate Professor, State University of New York - Upstate Medical University
Other Study IDs: 346301; R41MH111347 (NIH); R42MH111347 (NIH)
Record Dates: First submitted 2016-07-12; First posted 2016-07-14 (Estimated); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Autism Spectrum Disorder; Developmental Delay
Keywords: Autism; Asperger's Syndrome; microRNA; epigenetic; biomarker
MeSH Terms: conditions — Autism Spectrum Disorder; Learning Disabilities; Autistic Disorder; Asperger Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Salivary RNA
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- MCHAT-R Positive: Children identified at risk for the development of autism spectrum disorder (ASD) by scoring a 3 or higher on the MCHAT-R. Participants should not have a history of extreme pre-term birth or underlying neurological disorders such as seizures or cerebral palsy.
  Interventions: Other: Salivary collection; Other: Vineland Adaptive Behavior Scale-III Assessment; Other: Medical history questionaire; Other: Autism Diagnostic Observation Schedule -2nd edition (ADOS-2); Other: Mullen Scales of Early Learning

INTERVENTIONS:
Other: Salivary collection — Collection of saliva via swab for miRNA processing
Other: Vineland Adaptive Behavior Scale-III Assessment
Other: Medical history questionaire
Other: Autism Diagnostic Observation Schedule -2nd edition (ADOS-2)
Other: Mullen Scales of Early Learning

SUMMARY:
The goal of this study is to validate a panel of miRNAs that distinguish children with autism spectrum disorder (ASD) from their non-ASD peers with a positive MCHAT-R. These biomarkers may allow earlier diagnosis of autism, allowing earlier service, and also help us to understand some of the changes in the brains of autistic children.

DETAILED DESCRIPTION:
The central aim of this project is to validate a panel of expressed microRNA (miRNA) in the saliva of children identified at risk for developing ASD by the MCHAT-R. Further, this study aims to assess the value of the current panel as an adjunctive test that may increase specificity of MCHAT-R positive results, or affirm clinical diagnoses alongside the ADOS or other objective assessments.

The primary endpoints of this study are as follows:

1. Evaluate the diagnostic ability (sensitivity and specificity) of the current a salivary microtranscriptome panel for distinguishing children with ASD from their non-ASD peers.
2. Assess stability of the salivary microtranscriptome diagnosis over time, and interrogate longitudinal microtranscriptome levels relative to neuropsychological measures.

Secondary endpoints are the identification of microtranscriptome features whose concentrations correlate with ASD endophenotypes.

ELIGIBILITY:
Inclusion Criteria:

* Age at enrollment: 24 months to 48 months (inclusive)
* MCHAT-R score of 3 or greater
* Parent/guardian must be fluent in spoken English (required to complete study specific questionnaires etc)

Exclusion Criteria:

* confounding neurological (i.e. cerebral palsy, epilepsy), sensory (i.e. auditory or visual) impairments, and feeding tube dependence.
* history of extreme pre-term birth (< 32 weeks gestation)
* wards of the state
* Autistic subjects with known syndromic autism (attributed to a known genetic mutation)

Ages: 24 Months to 48 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study will compare salivary miRNA in children between the ages of 24 months and 48 months of age who are considered at risk for the development of autism spectrum disorder as identified by a score of 3 or greater on the MCHAT-R.
Sampling Method: Non-Probability Sample
Enrollment: 998 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Salivary miRNA profile | at the time of collect (from 18m to 6 years of age)
  Measures of miRNA abundance in saliva

SECONDARY OUTCOMES:
Measures of adaptive function | At time of enrollment (from 18m to 6 years of age)
  Vineland Adaptive Behavior Composite Score
Measures of early intellectual development | At time of enrollment (from 18m to 6 years of age)
  Mullen Scales of Early Learning
Measure of autistic behavior | At time of enrollment (from 18m to 6 years of age)
  Autism Diagnostic Observation Schedule (ADOS) Composite Score (Autism Group Only)

CONTACTS AND LOCATIONS:
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hicks SD, Ignacio C, Gentile K, Middleton FA. Salivary miRNA profiles identify children with autism spectrum disorder, correlate with adaptive behavior, and implicate ASD candidate genes involved in neurodevelopment. BMC Pediatr. 2016 Apr 22;16:52. doi: 10.1186/s12887-016-0586-x. PMID 27105825
- [Background] Hicks SD, Rajan AT, Wagner KE, Barns S, Carpenter RL, Middleton FA. Validation of a Salivary RNA Test for Childhood Autism Spectrum Disorder. Front Genet. 2018 Nov 9;9:534. doi: 10.3389/fgene.2018.00534. eCollection 2018. PMID 30473705
- [Derived] Hicks SD, Carpenter RL, Wagner KE, Pauley R, Barros M, Tierney-Aves C, Barns S, Greene CD, Middleton FA. Saliva MicroRNA Differentiates Children With Autism From Peers With Typical and Atypical Development. J Am Acad Child Adolesc Psychiatry. 2020 Feb;59(2):296-308. doi: 10.1016/j.jaac.2019.03.017. Epub 2019 Mar 27. PMID 30926572